CLINICAL TRIAL: NCT05359146
Title: Combined Beta- Plus Auger Electron Therapy Using a Novel Somatostatin Receptor Subtype 2 Antagonist Labelled With Terbium-161 (161Tb-DOTA-LM3): Beta Plus Study
Brief Title: Combined Beta- Plus Auger Electron Therapy Using a Novel Somatostatin Receptor Subtype 2 Antagonist Labelled With Terbium-161 (161Tb-DOTA-LM3)
Acronym: Beta plus
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: University Hospital, Basel, Switzerland (Other)
Collaborators: Swiss National Science Foundation (Other); Paul Scherrer Institute (PSI) (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 2022-00162; th21Wild
Record Dates: First submitted 2022-04-27; First posted 2022-05-03 (Actual); Last update posted 2024-04-19 (Actual); Status verified 2024-04

CONDITIONS: Neuroendocrine Neoplasia's (NENs); Gastroenteropancreatic Neuroendocrine Tumour (GEP-NET)
Keywords: Somatostatin receptor subtype 2 (SST2); 161Tb-DOTA-LM3; Somatostatin receptor subtype 2 (SST2) antagonist; Peptide receptor radionuclide therapy (PRRT); 177Lu-DOTATOC (177Lu-edotreotide); Auger electrons
MeSH Terms: conditions — Gastro-enteropancreatic neuroendocrine tumor | interventions — 177Lu-octreotide, DOTA(0)-Tyr(3)-

STUDY DESIGN:
Intervention Model Description: A randomized, cross-over, prospective, single-centre, open label phase 0 study, comparing the dosimetry of 177Lu-DOTATOC and 161Tb-DOTA-LM3 in the same patients.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Phase 0a, Group 1 (Experimental): The first test injection will be with 161Tb-DOTA-LM3; the second one will be with 177Lu-DOTATOC. The ~ 3 therapy cycles will be performed with 177Lu-DOTATOC.
  Test injection 1: 0.5 - 1 GBq ≤ 100 μg 161Tb-DOTA-LM3 with renal protection Test injection 2 (Cross over): 0.5 - 1 GBq ~ 200 μg 177Lu-DOTATOC with renal protection Not more than 6 weeks later patients will receive ~ 3 treatment cycles with 5.6 - 7.4 GBq 177Lu-DOTATOC in an interval of about 8 weeks (clinically established amount of activity). This is standard of care and not part of the study.
  Interventions: Drug: 161Tb-DOTA-LM3; Drug: 177Lu-DOTATOC
- Phase 0a, Group 2 (Experimental): The first test injection will be with 177Lu-DOTATOC; the second one will be with 161Tb-DOTA-LM3. The ~ 3 therapy cycles will be performed with 177Lu-DOTATOC.
  Test injection 1: Group 2: 0.5 - 1 GBq ~ 200 μg 177Lu-DOTATOC with renal protection Test injection 2 (Cross over): 0.5 - 1 GBq ≤ 100 μg 161Tb-DOTA-LM3 with renal protection Not more than 6 weeks later patients will receive ~ 3 treatment cycles with 5.6 - 7.4 GBq 177Lu-DOTATOC in an interval of about 8 weeks (clinically established amount of activity). This is standard of care and not part of the study.
  Interventions: Drug: 161Tb-DOTA-LM3; Drug: 177Lu-DOTATOC
- Phase 0b, Group 1 (Experimental): Both test injections will be with 161Tb-DOTA-LM3 (with different peptide amounts). The ~ 2 therapy cycles will be performed with 161Tb-DOTA-LM3.
  Test injection 1: ~ 2 GBq ≤ 100 μg 161Tb-DOTA-LM3 with renal protection Test injection 2: ~ 2 GBq ~ 300 μg 161Tb-DOTA-LM3 with renal protection Not more than 6 weeks later patients will receive ~ 2 cycles with ~ 3 GBq 161Tb-DOTA-LM3 in an interval of about 8 weeks if ~2 GBq is well tolerated
  Interventions: Drug: 161Tb-DOTA-LM3
- Phase 0b, Group 2 (Experimental): Start with the other peptide amount of 161Tb-DOTA-LM3. The ~ 2 therapy cycles will be performed with 161Tb-DOTA-LM3.
  Test injection 1: ~ 2 GBq ~ 300 μg 161Tb-DOTA-LM3 with renal protection Test injection 2: ~ 2 GBq ≤ 100 μg 161Tb-DOTA-LM3 with renal protection Not more than 6 weeks later patients will receive ~ 2 cycles with ~ 3 GBq 161Tb-DOTA-LM3 in an interval of about 8 weeks if ~2 GBq is well tolerated
  Interventions: Drug: 161Tb-DOTA-LM3

INTERVENTIONS:
Drug: 161Tb-DOTA-LM3 — 161Tb-DOTA-LM3 is a therapeutic medicinal product with three main components, namely (a) Terbium-161 (161Tb), a beta minus-, gamma- and Auger-/conversion electron-emitting radionuclide with a half-life of 6.96 days; (b) DOTA, a chelator that allows stable complexation of 161Tb; and (c) LM3, an antagonistic SST analogue which binds to SST2 receptors (SST2 receptor antagonist).
  All doses are presented as a sterile aqueous solution for i. v. infusion with renal protection.
Drug: 177Lu-DOTATOC — 177Lu-DOTATOC = 177Lu-edotreotide is a therapeutic medicinal product with three main components (a) Lutetium-177 (177Lu), a beta minus and gamma--emitting radionuclide with a half-life of 6.65 days; (b) DOTA, a chemical chelator that allows stable complexation of 177Lu; and (c) TOC (= [Tyr]3-octreotide) an agonistic somatostatin analogue which binds to SST2 and much less to SST5 receptors (SST2 receptor agonist).
  All doses are presented as a sterile aqueous solution for i. v. infusion with renal protection.
  Arms: Phase 0a, Group 1; Phase 0a, Group 2

SUMMARY:
The goal of this phase 0 proof-of concept study is to measure the therapeutic index (tumour to dose-limiting-organ dose ratios) of 161Tb-DOTA-LM3 in comparison to the current standard 177Lu-DOTATOC in the same gastroenteropancreatic neuroendocrine tumour (GEP-NET) patients in a randomized, cross-over design, in all patients.

Population to be studied are patients with diagnosed and metastasized secreting and non-secreting GEP-NEN (grade 1 and 2). The number of participants will be limited to 4 - 8 patients (phase 0a) and 4 - 8 patients (phase 0b). All patients will get the same treatment in a balanced cross-over order. The study will be divided into a phase 0a and phase 0b. Beforehand the selected patients will be randomised into two groups. In phase 0a one test injection with 161Tb-DOTA-LM3 and 177Lu-DOTATOC will administered in both randomised groups in a different order followed by ~ 3 cycles PRRT with 177Lu-DOTATOC in both groups. In phase 0b two test injections with 161Tb-DOTA-LM3 (with different peptide amounts) will administered in both randomised groups in a different order followed by ~2 cycles PRRT with 161Tb-DOTA-LM3 in both groups.

DETAILED DESCRIPTION:
Neuroendocrine neoplasia's (NENs) are a group of neoplasms arising from neuroendocrine cells and are most commonly found in the intestine, pancreas and lung. The overexpression of somatostatin receptor subtype 2 (SST2), is a characteristic of NENs and presents an important molecular target for the management of these tumours. Peptide receptor radionuclide therapy (PRRT) targets the SST2 through the administration of radiolabelled SST2 agonists such as 177Lu-DOTATOC and 177Lu-DOTATATE (Lutathera®). Although PRRT is one of the most efficient treatments for the management of NENs, it does only stabilize but not cure the disease. There is a need to improve PRRT with more effective radiopharmaceuticals. There is evidence that terbium-161 (161Tb) is more powerful that 177Lu not only in combination with SST2 agonists but particularly with SST2 antagonists.

The efficacy of PRRT can be enhanced by using a potent SST2 antagonist (DOTA-LM3) labelled with 161Tb. 161Tb-DOTA-LM3 has the following advantages compared to 177Lu-DOTATOC and 177Lu-DOTATATE: 1) SST2 antagonists bind to many more SST2-binding sites and accumulate mainly on the cellular membrane. 2) The Auger electrons of 161Tb deposit their high energy over a short distance (1-1000 nm) resulting in a high relative biological effectiveness mainly to the cell membrane which seems to be more radiosensitive than the cytoplasm. 161Tb-DOTA-LM3 does, therefore, not only deliver dose by β- radiation, but also through the emission of conversion and Auger electrons which leads to a 3 - 4 fold increased dose to single cancer cells compared to 177Lu-DOTA-LM3.

The goal of this phase 0 proof-of concept study is to measure the therapeutic index (tumour to dose-limiting-organ dose ratios) of 161Tb-DOTA-LM3 in comparison to the current standard 177Lu-DOTATOC in the same gastroenteropancreatic neuroendocrine tumour (GEP-NET) patients.

ELIGIBILITY:
Inclusion Criteria:

* Written consent
* Patients with diagnosed and metastasized secreting and non-secreting GEP-NEN (grade 1 and 2)
* Absence of a curative surgical option
* At least 2 measurable tumours based on RECIST 1.1 (minimal tumour diameter of 1 cm)
* Documentation of a positive 68Ga-DOTATOC/-TATE positron emission tomography (PET)/CT (in vivo detection of SST2 on GEP-NENs)
* Indication for PRRT
* Patient of any gender and of age older than 18
* Female patients of child-bearing age (who are not surgically sterilized or are less than 2 years in their menopause) must use a medically accepted contraceptive and must agree to use it during and till 3 months after the treatment. As acceptable contraceptive count sexual abstinence or double contraceptive methods: hormonal contraceptive (oral, transdermal, implants or injections) in combination with barrier methods (spiral, condom, diaphragm)
* Eastern Cooperative Oncology Group (ECOG) ≤ 2
* Blood parameters:

  h) Leucocytes ≥ 3*109/L i) Haemoglobin ≥ 90 g/L j) Thrombocytes ≥ 90*109/L k) Estimated glomerular filtration rate ≥ 50 ml/min or Creatinine < 150 μmol/l l) Albumin > 25 g/L m) alanine aminotransferase (ALT), aspartate aminotransferase (AST), alkaline phosphatase (AP): ≤ 5 times upper standard value n) Bilirubin ≤ 2 times upper standard value

Exclusion Criteria:

* Known intolerance against 177Lu, 161Tb, DOTA, TOC, LM3, SST analogues or against one of the components of 177Lu-DOTATOC or 161Tb-DOTA-LM3
* Bone/bone marrow metastases located in the lumbar spine if they affect the bone marrow dose estimation
* Ongoing infection at the screening visit or a serious infection in the past 4 weeks
* Administration of another investigational product in the last 60 days before Visit 1 Day 1
* Prior or planed administration of a therapeutic radio-pharmaceutical during 8 half-lives of the used radio-pharmaceutical's radionuclide, also during the ongoing study
* Any extensive radiotherapy involving bone marrow over the last 3 months before inclusion to the study
* Chemotherapy in the last 4 weeks before inclusion
* Pregnant or breastfeeding female patients. A pregnancy test will be performed in all women of child-bearing age.
* Any uncontrolled significant medical, psychiatric or surgical condition (active infection, unstable angina pectoris, cardiac arrhythmia, poorly controlled hypertension, poorly controlled diabetes mellitus [HbA1c ≥ 9%], uncontrolled congestive heart disease, etc.) or laboratory findings that might jeopardize the patient's safety or that would limit compliance with the objectives and assessments of the study. Any mental conditions which prevent the patient from understanding the type, extent and possible consequences of the study and/or an uncooperative attitude from the patient.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Estimated)
Dates: Start 2023-03-28 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Change in bone marrow doses after sequential injection of a non-therapeutic test activity of 161Tb-DOTA-LM3 and 177Lu-DOTATOC in the same patients. | ~ 3, ~ 24, ~ 72 and ~ 168 hours post injection
  Assessment and comparison of the tumour-to-bone marrow dose ratio of 161Tb-DOTA-LM3 vs 177Lu-DOTATOC. In order to get kinetic information of 161Tb-DOTA-LM3 and 177Lu-DOTATOC for this task total body scintigraphy and SPECT/CT of abdomen are performed at different time points post injection 161Tb-DOTA-LM3 or 177Lu-DOTATOC: ~ 3, ~ 24, ~ 72 and ~ 168 hours.
Change in kidney doses after sequential injection of a non-therapeutic test activity of 161Tb-DOTA-LM3 and 177Lu-DOTATOC in the same patients. | ~ 3, ~ 24, ~ 72 and ~ 168 hours post injection
  Assessment and comparison of the tumour-to-kidney dose ratio of 161Tb-DOTA-LM3 vs 177Lu-DOTATOC. In order to get kinetic information of 161Tb-DOTA-LM3 and 177Lu-DOTATOC for this task total body scintigraphy and SPECT/CT of abdomen are performed at different time points post injection 161Tb-DOTA-LM3 or 177Lu-DOTATOC: ~ 3, ~ 24, ~ 72 and ~ 168 hours.

SECONDARY OUTCOMES:
Change in median tumour dose per gigabequerel (GBq) injected activity | ~ 3, ~ 24, ~ 72 and ~ 168 hours post injection
  Assessment of the median tumour dose per GBq injected activity (Median of the mean of 2 - 6 tumours per patient which can be identified with both compounds.). Kinetic information of the biodistribution of 161Tb-DOTA-LM3 and 177Lu-DOTATOC for dosimetry calculations will be generated by performing sequential SPECT/CT scans for example at ~ 3, ~ 24, ~ 72 and ~ 168 hours.
Change in median tumour-to-bone marrow- dose ratio | ~ 3, ~ 24, ~ 72 and ~ 168 hours post injection
  Kinetic information of the biodistribution of 161Tb-DOTA-LM3 and 177Lu-DOTATOC for dosimetry calculations will be generated by performing sequential SPECT/CT scans for example at ~ 3, ~ 24, ~ 72 and ~ 168 hours.
Change in median tumour-to-kidney- dose ratio | ~ 3, ~ 24, ~ 72 and ~ 168 hours post injection
  Kinetic information of the biodistribution of 161Tb-DOTA-LM3 and 177Lu-DOTATOC for dosimetry calculations will be generated by performing sequential SPECT/CT scans for example at ~ 3, ~ 24, ~ 72 and ~ 168 hours.
Bone marrow toxicity using the Common Terminology Criteria for Adverse Events (CTCAE) version 5.0. | ~ 3, ~ 24, ~ 72 and ~ 168 hours post injection
  Assessment of bone marrow toxicity after test injection of 177Lu-DOTATOC and 161Tb-DOTA-LM3 using the Common Terminology Criteria for Adverse Events (CTCAE) version 5.0.
Change in median dose per GBq injected activity in other organs than bone marrow and kidneys | ~ 3, ~ 24, ~ 72 and ~ 168 hours post injection
  Assessment of the median dose per GBq injected activity in other organs than bone marrow and kidneys. Kinetic information of the biodistribution of 161Tb-DOTA-LM3 and 177Lu-DOTATOC for dosimetry calculations will be generated by performing sequential SPECT/CT scans for example at ~ 3, ~ 24, ~ 72 and ~ 168 hours.

CONTACTS AND LOCATIONS:
Overall Officials: Damian Wild, Prof. Dr. med., Study Director — Division of Nuclear Medicine, University Hospital Basel
Locations (1):
- Division of Nuclear Medicine, University Hospital Basel, Basel, Switzerland